CLINICAL TRIAL: NCT04075500
Title: Optimal Detection of Atrial Fibrillation in Transient Ischemic Attack
Brief Title: Optimal Detection of Atrial Fibrillation in TIA
Acronym: ODEA-TIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alfried Krupp Krankenhaus (Other)
Collaborators: Medtronic Bakken Research (Industry); Coordinating Centre for Clinical Trials Heidelberg (Unknown); Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AKKNeuro2019July
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation; Transient Ischemic Attack
Keywords: atrial fibrillation; monitoring; ECG; ischemic attack
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Attack, Transient | interventions — Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Patient will be randomized to either receive 24-h Holter Monitoring or receive one of the two modes for prolonged ECG recording (interventional arms). Patient will either undergo 28-day ECG recording using a commercially available Holter Recorder that can function as a non-invasive ECG patch or receive an implantable cardiac device (REVEAL LINQ).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (No Intervention): Control arm, 24-h Holter monitoring
- Arm 2 (Other): 1st interventional arm, subcutaneously implanted event recorder (REVEAL LINQ)
  Interventions: Device: Subcutaneously implanted event recorder (REVEAL LINQ)
- Arm 3 (Other): 2nd interventional arm, 28-day continuous ECG monitoring
  Interventions: Device: 28-day non-invasive continuous ECG monitoring (patch)

INTERVENTIONS:
Device: Subcutaneously implanted event recorder (REVEAL LINQ) — Patients receive a subcutaneously implantable cardiac device (REVEAL LINQ).
  Arms: Arm 2
Device: 28-day non-invasive continuous ECG monitoring (patch) — Patients receive a non-invasive continuous ECG monitoring (patch)
  Arms: Arm 3

SUMMARY:
Transient ischemic attack (TIA) is a common neurologic emergency. Although the detection of atrial fibrillation (AF) has identical consequences for preventive therapy in patients with ischemic stroke and TIA, the management setting and diagnostic pathways frequently differ substantially between both manifestations. Despite these differences between stroke and TIA patients, previous studies have investigated diagnostic work-up for AF primarily in stroke patients. Thus, there is no common practice or "gold standard" of rhythm monitoring for TIA patients in most healthcare systems and the optimal method and duration of cardiac monitoring for TIA patients is currently unknown. This is likely to result in a substantial under-diagnosis of AF in TIA patients, failure to initiate appropriate secondary preventive medication (i.e. anticoagulation) and ultimately the occurrence of many otherwise preventable strokes.

The primary research question of the trial is whether prolonged ECG recording using a subcutaneously implanted event recorder increases the detection rate of paroxysmal AF (pAF) within 6 months after the event in patients with recent TIA both compared to 24-h ECG recording and compared to prolonged ECG recording using non-invasive continuous ECG recording for 28 days AND To determine whether 28-day non-invasive ECG monitoring increases the detection rate of pAF within 6 months after the event compared to 24-h ECG recording.

DETAILED DESCRIPTION:
Transient ischemic attacks (TIA) are a common neurologic emergency. Clinical management guidelines recommend oral anticoagulation for TIA patients suffering from atrial fibrillation (AF). Therefore, a diagnosis of AF in TIA patients has a major impact on the choice of adequate secondary stroke prevention. However, detection of paroxysmal AF in patients with TIA can be challenging. AF remains undetected in a relevant proportion of stroke and TIA patients using current routine diagnostic procedures. The actual prevalence of AF in TIA patients is unknown.

Although the detection of AF has identical consequences for preventive therapy in patients with ischemic stroke and TIA, the management setting and diagnostic pathways frequently differ substantially between both manifestations. So far, only limited data exist on AF detection after TIA specifically, and the best method for diagnosis of AF has not been established. The usefulness of prolonged rhythm monitoring using event recorders or non-invasive continuous ECG in TIA patients has not been determined. While the use of an AF detection tool in TIA patients is desirable, an adequate use of resources of AF detection technologies in unselected TIA patients may be needed for this large scale health care problem. Identifying TIA patients that are at increased risk of suffering from AF using clinical and blood-based biomarkers and therefore most likely to benefit from such diagnostic procedures would be useful.

The primary research question of the trial is whether prolonged ECG recording using a subcutaneously implanted event recorder increases the detection rate of paroxysmal AF (pAF) within 6 months after the event in patients with recent TIA both compared to 24-h ECG recording and compared to prolonged ECG recording using non-invasive continuous ECG recording for 28 days AND To determine whether 28-day non-invasive ECG monitoring increases the detection rate of pAF within 6 months after the event compared to 24-h ECG recording. The ODEA-TIA trial is an investigator initiated prospective, multicentre, randomized, open study with blinded outcome assessment comparing different diagnostic methods for detection of paroxysmal AF in patients with recent TIA. The primary endpoint is the rate of AF detection during the 6 months after randomization. Approximately 40 centers in Europe (Germany and Spain) will participate in this trial. Patients with a recent TIA fulfilling the eligibility criteria (see below) will be randomized in a 1:1:1 fashion between 24 h arrhythmia monitoring (control arm) and the two procedures for prolonged ECG monitoring (interventional arms). That means we have two interventional arms, patients receiving either continuous 28d non-invasive ECG monitoring or ECG event recording using a subcutaneously implanted event recorder.

ELIGIBILITY:
Eligibility Criteria:

Study Population Patients with a recent TIA will be enrolled during a period of approximately 24 months at participating European stroke centres. TIA patients may be enrolled after initial management as inpatients or outpatients. Consecutive screening and enrolment will be strongly encouraged and a screening log will be implemented at each site.

Inclusion Criteria

* Written informed consent by patient.
* Age ≥ 50 years.
* TIA diagnosed by a stroke physician defined as rapidly developing clinical signs of focal or global disturbances of cerebral function, lasting less than 24 hours with no apparent non-vascular cause
* 12-channel ECG available before enrolment
* Brain imaging available before enrolment (CCT or cranial MRI)
* Vascular imaging of cervical vessels performed
* Enrolment within 28 days after TIA episode. Exclusion Criteria
* Previously documented history of AF
* Ischemic stroke within the last 6 months before enrolment
* Pre-screening monitoring for cardiac arrhythmias lasting ≥72 hours
* AF lasting > 30 s on a 12 channel ECG or other ECG recording technique prior to enrolment
* Life expectancy less than 1 year.
* Significant stenosis > 50% in intracranial or extracranial vessels which, in the opinion of the investigator, is the likely cause of the patients TIA.
* Severely disabled patients (i.e. modified Rankin Score >3)
* Lack of therapeutic consequence in case of diagnosis of AF (e.g. other indication for long term anticoagulation
* Pacemaker or Implanted Cardiac Defibrillator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of newly detected AF at 6 month after study enrolment in patients with recent TIA | 6 month
  Self reported or by other means detected newly AF

SECONDARY OUTCOMES:
Prevalence of AF in TIA patients as determined by prolongend ECG Monitoring techniques | 24 month
  Self reported or by other means detected newly AF
Rate of newly detected AF at 12 and 24 month after study enrolment in patients with recent TIA | 12 and 24 month
  Self reported or by other means detected newly AF in longterm ECG Monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Roland Veltkamp, MD, Principal Investigator — Initiator of study, leader PI
Locations (27):
- Germany (16):
  - Universitätsklinikum Aachen, Neurologie, Aachen
  - Rhön Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale
  - Vivantes Klinikum Neukölln, Berlin
  - Carl-Thiem-Klinikum Cottbus; Klinik für Neurologie, Cottbus
  - Klinikum Dortmund, Klinikzentrum Mitte / Neurologie, Dortmund
  - Alfried Krupp Krankenhaus, Essen
  - Universitätsmedizin Frankfurt; Klinik für Neurologie;, Frankfurt
  - Bezirkskliniken Schwaben; Bezirkskrankenhaus Günzburg; Klinik für Neurologie, Günzburg
  - Krankenhaus Marth-Maria-Halle-Dölau GmbH; Klinik für Neurologie, Halle
  - Universitätsmedizin Halle; Universitätsklinikum Halle (Saale); Klinik und Poliklinik für Neurologie, Halle
  - Universitätsklinik Heidelberg, Neurologie, Heidelberg
  - Universität Leipzig, Medizinische Fakultät; Klinik und Poliklinik für Neurologie, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Tübingen; Neurologische Universitätsklinik; Abt. Neurologie mit Schwerpunkt vaskuläre Erkrankungen, Tübingen
  - RKU Universitäts- und Rehabilitationskliniken Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Spain (11):
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Dr. Josep Trueta, Girona
  - Complejo Hospitalario Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No